CLINICAL TRIAL: NCT02394938
Title: A Randomized Controlled Trial of Listen Recorded Music for Hearth Failure Patients
Brief Title: Effects of Recorded Music in Heart Failure Patients
Acronym: EMSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Principal Investigator, CARLO DESCOVICH, MD, Azienda Usl di Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE 14123
Record Dates: First submitted 2015-02-17; First posted 2015-03-20 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Heart Diseases
Keywords: Music therapy
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MUSIC (Experimental): In addition to the standard care, heart failure patients assigned to the music group will listen recorded classical music.
  Interventions: Other: MUSIC
- CONTROL (No Intervention): Heart Failure patients assigned to the control group will receive standard care only. The standard care will consist in nursing and medical counselling, self-care education and medication.

INTERVENTIONS:
Other: MUSIC — In addition to the standard care,patients assigned to the music group will listen recorded classical music. Music will be delivered with a mp3 Player and headphones Music will be listened by the patient in his home.The music play list will be formed by a classical repertoire.During the intervention patients will be recommended to listen to the music for 3 months. Also patients will be asked to listen to the music once or more than once per day, at any time, for a total of 30 minutes per day.Music will be listen at 50-60 decibels below the threshold of 85 db established for listening to portable media devices such as compact disc and MP3 players.Music in this protocol will have a tempo/rhythm in a range of 60-80 beats per minute (bpm).
  Arms: MUSIC

SUMMARY:
Aims. To describe a new conceptual framework and to test the effectiveness of a recorded music listening protocol on symptom burden and quality of life in heart failure patients.

DETAILED DESCRIPTION:
Background. Heart failure is an important public health problem. Many heart failure patients experience symptoms burden and poor quality of life, even after the improvements in pharmacological treatments. Recorded music listening was shown to improve outcomes in cardiovascular patients but it was never tested on heart failure patients. Methods. This study is a multi-centred single-blind randomized controlled trial that will involve 150 patients. Eligible patients will have a diagnosis of heart failure, in New York Hearth Association functional classification I to III, and will be recruited from seven outpatient clinics in Northern Italy. Patients will be randomly allocated in a 1:1 ratio to receive the recorded music listening intervention or the standard care for 3 months. Data will be collected at baseline and first, second and three month during the intervention, and at six month for follow-up. The following variables will be collected from heart failure patients by validated outcome measuring instruments for quality of life (primary endpoint), use of emergency services, re-hospitalization rates, all-cause mortality,self-care, somatic symptoms, quality of sleep ,anxiety and depression, cognitive state. The study has been funded by Italian Heart Failure Association in November 2014 with number 01/04. Ethical approval was gained in December 22, 2015.

Discussion. This study will be a trial to examine the effect of recorded music listening on heart failure patients and will inform clinical practice and will provide empirical data for a new music protocol intervention evidence based. The new framework may be helpful for future research focused on music effect in heart failure patients.

Sample size calculation.The sample size will be based on the primary endpoint of quality of life measured with the Minnesota Living with Heart Failure Questionnaire. Considering two balanced groups (n1 = n2), a medium effect size (d = 0.5), α error of 5% and power of 80% to detect differences between groups, it would be necessary to enrol a total of 128 (n1 = n2 = 64) patients. A medium effect size d = 0.5 implies a sample different expectation of 10 points at the Minnesota Living with Heart Failure Questionnaire, in according to study of Parati and colleges (Parati, Malfatto et al. 2008). Given the ordinal nature of the variable, and assuming a normal distribution of scores, to maintain power to the expected value (80%), we should multiply by π / 3 (asymptotic relative efficiency value), obtaining a total of 134 subjects. Finally, assuming a drop-out of 10% for group (Park, Park et al. 2012), it will needed to enrol a total of 150 patients, 75 subjects per group. Data analysis.

Data from patients will entered into spreadsheet files and checked for data errors independently by another researcher. Analyses will conducted using SPSS 19.0 (IBM Corporation, Armonk,NY). Descriptive statistics, mean, standard deviation, frequencies, median and interquartile ranges will be used to describe scale scores and social-demographic and clinical data. All tests will be two-tailed. A probability value <0.05 will be considered the minimum level of statistical significance. To test the means differences between groups at baseline and at 1st 2nd, 3th month and at 6th month after enrolment, repeated measures ANOVA with Bonferroni post-hoc test will be used. If repeated measures ANOVA will show an effect of treatment, MANCOVA analysis will be used to verify possible association between the outcome and continuous predictor variables. To calculate the correlations between the scores of the different questionnaires the correlation coefficient of Pearson or Spearman will used with. Fisher's exact test or χ2 test will be used to identify differences in use of emergency services, hospitalization and mortality between intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of heart failure according to the guidelines specified by the European Society of Cardiology ;
* NYHA functional classification I to III, including patients with preserved ejection fraction (HFPEF) and with a reduced ejection fraction (HFREF);
* the presence of a formal or informal caregiver;
* signed informed consent.

Exclusion Criteria:

* deafness ;
* severe neurological disorder (Parkinson, multiple sclerosis, Alzheimer's disease;
* severe psychiatric disorder;
* frank dementia,
* reduced level of consciousness.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in heart failure specific quality of life (Minnesota Living with Heart Failure Questionnaire) | Baseline, 1st 2nd, 3th, 6th month
  The heart failure specific quality of life will be measured with the Minnesota Living with Heart Failure Questionnaire.

SECONDARY OUTCOMES:
Use of emergency services | 1st, 2nd, 3th, 6th month
Generic quality of life (measured with the Short Form -12.) | Baseline, 1st 2nd, 3th, 6th month
  The generic quality of life will be measured with the Short Form -12.
Self-care (Self-Care of Heart Failure Index version 6.2) | Baseline, 1st 2nd, 3th, 6th month
  Patient's self-care will be measured with the Self-Care of Heart Failure Index version 6.2
Somatic perception of heart failure symptoms (Heart Failure Somatic Perception Scale) | Baseline, 1st 2nd, 3th, 6th month
  Somatic perception of heart failure symptoms. They will be evaluated with the Heart Failure Somatic Perception Scale
Sleep quality (Pittsburgh Sleep Quality Index) | Baseline, 1st 2nd, 3th, 6th month
  Sleep quality. Sleep quality will be measured with the Pittsburgh Sleep Quality Index
Anxiety and depression (Hospital Anxiety and Depression Scale) | Baseline, 1st 2nd, 3th, 6th month
  Anxiety and depression will be measured with the
Cognition (Montreal Cognitive Assessment) | Baseline, 1st 2nd, 3th, 6th month
  Cognition will be measured by Montreal Cognitive Assessment
Hospitalization | 1st, 2nd, 3th, 6th month
Mortality | 1st, 2nd, 3th, 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Pirazzini, MSN, Principal Investigator — AUSL Bologna
Locations (1):
- Francesco Burrai, Bologna, Bologna, Italy

REFERENCES:
- [Result] Bernardi L, Porta C, Casucci G, Balsamo R, Bernardi NF, Fogari R, Sleight P. Dynamic interactions between musical, cardiovascular, and cerebral rhythms in humans. Circulation. 2009 Jun 30;119(25):3171-80. doi: 10.1161/circulationaha.108.806174. PMID 19569263
- [Result] Chanda ML, Levitin DJ. The neurochemistry of music. Trends Cogn Sci. 2013 Apr;17(4):179-93. doi: 10.1016/j.tics.2013.02.007. PMID 23541122
- [Result] Fancourt D, Ockelford A, Belai A. The psychoneuroimmunological effects of music: a systematic review and a new model. Brain Behav Immun. 2014 Feb;36:15-26. doi: 10.1016/j.bbi.2013.10.014. Epub 2013 Oct 21. PMID 24157429
- [Result] Hanser SB. Music therapy in cardiac health care: current issues in research. Cardiol Rev. 2014 Jan-Feb;22(1):37-42. doi: 10.1097/CRD.0b013e318291c5fc. PMID 23535529
- [Result] Mandel SE, Hanser SB, Secic M, Davis BA. Effects of music therapy on health-related outcomes in cardiac rehabilitation: a randomized controlled trial. J Music Ther. 2007 Fall;44(3):176-97. doi: 10.1093/jmt/44.3.176. PMID 17645384
- [Result] Trappe HJ. The effects of music on the cardiovascular system and cardiovascular health. Heart. 2010 Dec;96(23):1868-71. doi: 10.1136/hrt.2010.209858. PMID 21062776
- [Derived] Burrai F, Hasan W, Fancourt D, Luppi M, Di Somma S. A Randomized Controlled Trial of Listening to Recorded Music for Heart Failure Patients: Study Protocol. Holist Nurs Pract. 2016 Mar-Apr;30(2):102-15. doi: 10.1097/HNP.0000000000000135. PMID 26871248